CLINICAL TRIAL: NCT01637311
Title: Peroral Endoscopic Remyotomy for Failed Heller Myotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSNJ-POEM
Record Dates: First submitted 2012-07-03; First posted 2012-07-11 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-05

CONDITIONS: Esophageal Achalasia
Keywords: Peroral endoscopic myotomy; Heller myotomy; persistent/recurrent achalasia.
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Failed HM (Experimental): Patients were eligible for enrollment in the study if they were age greater than 18 years and had recurrence/persistence of symptoms after primary HM with an Eckardt symptom score ≥ 4.
  Interventions: Procedure: POEM

INTERVENTIONS:
Procedure: POEM — Peroral endoscopic myotomy (POEM) has recently been described as a new minimally invasive endoscopic myotomy technique intending a permanent cure from primary achalasia.

SUMMARY:
Achalasia is a rare esophageal motility disorder, which is characterized clinically by symptoms of dysphagia, regurgitation, weight loss and chest pain. With respect to long-term efficacy, Heller myotomy (HM) using an open or a laparoscopic approach has gained wide acceptance as the procedure of choice for the management of patients with primary achalasia in recent years. Although good or excellent long-term symptomatic response rates can be achieved in more than 90% of patients undergoing HM, recurrence or persistence of symptoms occurs in approximately 20%. Controversy exists regarding the therapy of patients with failed success after HM. Peroral endoscopic myotomy (POEM) has recently been described as a new minimally invasive endoscopic myotomy technique intending a permanent cure from primary achalasia. Our purpose was to evaluate the efficacy and the feasibility of POEM for patients with failed HM.

DETAILED DESCRIPTION:
1. Patients were eligible for enrollment in the study if they were age greater than 18 years and had recurrence/persistence of symptoms after primary HM with an Eckardt symptom score ≥ 4. The diagnosis of achalasia was made on the basis of the absence of peristalsis and on impaired relaxation of the LES on established methods (barium swallow, manometry, esophagogastroduodenoscopy (EGD)). Exclusion criteria were severe cardiopulmonary disease or other serious disease leading to unacceptable surgical risk, pseudoachalasia, and megaesophagus (diameter of > 7 cm).
2. All patients were scheduled for a follow-up visit at 1 month after POEM for EGD and manometry. Symptoms were assessed 1 month after treatment in the clinic and every 3 months thereafter via telephone questionnaires.
3. The primary outcome of the study was therapeutic success (a reduction in the Eckardt score to ≤3) at the follow-up assessment. The secondary outcomes included procedure-related adverse events, LES pressure on manometry pre- and post POEM, reflux symptoms and medication use before and after POEM, and procedure-related parameters such as procedure time, hospital stay, and myotomy length.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Recurrence/persistence of symptoms after primary HM with an Eckardt symptom score ≥ 4
* The diagnosis of achalasia was made on the basis of the absence of peristalsis and on impaired relaxation of the LES on established methods (barium swallow, manometry, esophagogastroduodenoscopy)

Exclusion Criteria:

* Severe cardiopulmonary disease or other serious disease leading to unacceptable surgical risk
* Pseudoachalasia
* megaesophagus (diameter of > 7 cm)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Therapeutic success (a reduction in the Eckardt score to ≤3) | Symptoms were assessed 1 month after treatment in the clinic and every 3 months thereafter via telephone questionnaires.

SECONDARY OUTCOMES:
Procedure-related adverse events | All patients were scheduled for a follow-up visit at 1 month after POEM for EGD.
Lower esophageal sphincter (LES) pressure on manometry | All patients were scheduled for a follow-up visit at 1 month after POEM for EGD and manometry
Reflux symptoms and medication use before and after POEM | Symptoms were assessed 1 month after treatment in the clinic and every 3 months thereafter via telephone questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Hong Zhou, MD,PhD, Study Director — Endoscopy Center and Endoscopy Research Institute, Zhongshan Hospital, Fudan University, Shanghai, China
Locations (1):
- Endoscopy Center and Endoscopy Research Institute, Zhongshan Hospital, Fudan University, Shanghai, China

REFERENCES:
- [Background] Eckardt AJ, Eckardt VF. Treatment and surveillance strategies in achalasia: an update. Nat Rev Gastroenterol Hepatol. 2011 Jun;8(6):311-9. doi: 10.1038/nrgastro.2011.68. Epub 2011 Apr 26. PMID 21522116
- [Background] Zaninotto G, Costantini M, Portale G, Battaglia G, Molena D, Carta A, Costantino M, Nicoletti L, Ancona E. Etiology, diagnosis, and treatment of failures after laparoscopic Heller myotomy for achalasia. Ann Surg. 2002 Feb;235(2):186-92. doi: 10.1097/00000658-200202000-00005. PMID 11807357
- [Background] Gockel I, Junginger T, Eckardt VF. Persistent and recurrent achalasia after Heller myotomy: analysis of different patterns and long-term results of reoperation. Arch Surg. 2007 Nov;142(11):1093-7. doi: 10.1001/archsurg.142.11.1093. PMID 18025339
- [Result] Iqbal A, Tierney B, Haider M, Salinas VK, Karu A, Turaga KK, Mittal SK, Filipi CJ. Laparoscopic re-operation for failed Heller myotomy. Dis Esophagus. 2006;19(3):193-9. doi: 10.1111/j.1442-2050.2006.00564.x. PMID 16722998
- [Result] Duffy PE, Awad ZT, Filipi CJ. The laparoscopic reoperation of failed Heller myotomy. Surg Endosc. 2003 Jul;17(7):1046-9. doi: 10.1007/s00464-002-8570-y. Epub 2003 May 7. PMID 12730729
- [Result] Rakita S, Villadolid D, Kalipersad C, Thometz D, Rosemurgy A. Outcomes promote reoperative Heller myotomy for symptoms of achalasia. Surg Endosc. 2007 Oct;21(10):1709-14. doi: 10.1007/s00464-007-9226-8. Epub 2007 Apr 14. PMID 17440784
- [Result] Inoue H, Minami H, Kobayashi Y, Sato Y, Kaga M, Suzuki M, Satodate H, Odaka N, Itoh H, Kudo S. Peroral endoscopic myotomy (POEM) for esophageal achalasia. Endoscopy. 2010 Apr;42(4):265-71. doi: 10.1055/s-0029-1244080. Epub 2010 Mar 30. PMID 20354937
- [Result] von Renteln D, Inoue H, Minami H, Werner YB, Pace A, Kersten JF, Much CC, Schachschal G, Mann O, Keller J, Fuchs KH, Rosch T. Peroral endoscopic myotomy for the treatment of achalasia: a prospective single center study. Am J Gastroenterol. 2012 Mar;107(3):411-7. doi: 10.1038/ajg.2011.388. Epub 2011 Nov 8. PMID 22068665
- [Result] Ren Z, Zhong Y, Zhou P, Xu M, Cai M, Li L, Shi Q, Yao L. Perioperative management and treatment for complications during and after peroral endoscopic myotomy (POEM) for esophageal achalasia (EA) (data from 119 cases). Surg Endosc. 2012 Nov;26(11):3267-72. doi: 10.1007/s00464-012-2336-y. Epub 2012 May 19. PMID 22609984